CLINICAL TRIAL: NCT00381368
Title: Phase II Open Label Study to Establish the Safety and Efficacy of Intravenous Loading Dose of Ibandronate 6 mg in 3 Consecutive Days in Breast Cancer Patients With Skeletal Metastases
Brief Title: Safety and Efficacy Study of Intravenous Loading Dose of Ibandronate in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20115; EudraCT: 2006-000697-74
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; skeletal metastases; bisphosphonate therapy; Breast cancer with painful skeletal metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — Ibandronic Acid

INTERVENTIONS:
Drug: Ibandronic acid

SUMMARY:
The purpose of the study is to determine the efficacy and safety of a three time repeated loading dose of intravenous ibandronate (ibandronic acid), 6 mg, in breast cancer patients with painful skeletal metastases.

DETAILED DESCRIPTION:
Painful skeletal metastases are a common site of advanced disease. For instance, in breast cancer, and despite cancer treatments (radiotherapy, cytotoxic treatment and adequate treatment of pain), the patients often need additional treatments that may relieve their symptoms. Bisphosphonates, such as ibandronic acid, have in pilot studies shown a significant decrease in pain scores, both after loading dose and after long-term treatment. In this study the safety and efficacy of an intravenous loading dose of three times 6 mg ibandronate during three consecutive days in breast cancer patients with painful skeletal metastases will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer with presence of bone metastases
* Pain score over 4 on the VAS

Exclusion Criteria:

* Patients with pathological fractures or medulla compression or neuropathic pain
* Patients with infection or corticosteroid treatment
* Pregnant or lactating patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2006-10

PRIMARY OUTCOMES:
Worst and average pain in movement and rest on the visual analogue scale (VAS) before the first dose, on days 2, 3, 7 and on day 28
Analgesic consumption during the same period will additionally be assessed

SECONDARY OUTCOMES:
Bone markers: serum 1CTP, serum P1NP, serum NTX on day 1 before dosing, and on days 7 and 28
World Health Organization (WHO) performance status
Safety: serum cystatin C and serum creatinine, and reporting of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Outi Paija, MD, PhD, Principal Investigator — Dept of Oncology, Turku University Hospital, Finland
Locations (3):
- Finland (3):
  - Dept of Oncology, Helsinki University Central Hospital, Helsinki, Helsinki
  - Dept of Oncology, Oulu University Hospital, Oulu, Oulu
  - Dept of Oncology, Tampere University Hospital, Tampere